CLINICAL TRIAL: NCT06734741
Title: Prospective Clinical Evaluation of COVID/Flu Detect™ Rapid Self-Test in Symptomatic Subjects for Non-Prescription Over-the-Counter (OTC) Use
Status: Completed | Type: Observational
Sponsor: InBios International, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: COVID-FLU-OTC 2024; W81XWH-20-F-0253 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2024-12-10; First posted 2024-12-16 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: COVID-19; Influenza A; Influenza B
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal swab sample in transport medium collected from study participant by a healthcare provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: COVID/Flu Detect™ Rapid Self-Test — The COVID/Flu Detect™ Rapid Self-Test is an investigational qualitative lateral flow immunoassay designed for the detection and differentiation of SARS-CoV-2, influenza A, and influenza B protein antigens in nasal swab samples. It is intended for non-prescription over-the-counter (OTC) use.

SUMMARY:
The goal of this study is to evaluate the performance of the COVID/Flu Detect™ Rapid Self-Test when used in a home-like setting by lay users. The COVID/Flu Detect™ Rapid Self-Test is an investigational device intended for the qualitative detection and differentiation of SARS-CoV-2, influenza A, and influenza B protein antigens in nasal swab samples. Participants who are aged two (2) years and older and have symptoms of respiratory illness consistent with SARS-CoV-2 and influenza infection may be enrolled. Participants will use the COVID/Flu Detect™ Rapid Self-Test to self-collect, self-test, and interpret the results. Participants will have a nasal swab sample collected by a healthcare provider for comparator testing by PCR tests for SARS-CoV-2, influenza A, and influenza B. Researchers will compare the results of the COVID/Flu Detect™ Rapid Self-Test obtained by the participants to results from the PCR comparator tests to evaluate performance.

DETAILED DESCRIPTION:
This study will be a multi-site, all-comers, clinical trial assessing the positive percent agreement (PPA) and negative percent agreement (NPA) of the COVID/Flu Detect™ Rapid Self-Test, an investigational qualitative lateral flow immunoassay intended for non-prescription over-the-counter (OTC) use. Participants who are aged 2 years and older and meet the eligibility criteria will be enrolled for testing on the COVID/Flu Detect™ Rapid Self-Test and for comparator testing on (1) an FDA-cleared or emergency use authorized (EUA) SARS-CoV-2 RT-PCR test, (2) an FDA-cleared influenza A RT-PCR test, and (3) an FDA-cleared influenza B RT-PCR test.

After obtaining informed consent, participants' age, sex, days post-symptom onset, signs and symptoms of respiratory illness, comorbidities, any medications taken or administered, influenza/COVID-19 vaccination history, race/ethnicity, socioeconomic status, and educational background will be collected. Next, two (2) anterior nasal swab samples will be collected from each participant, with at least a 15-minute normalization period between swab sample collections. One (1) of the nasal swab samples will be collected by a healthcare provider (HCP) from the participant. This nasal swab sample will be sent for comparator testing. The other nasal swab sample will be self-collected or collected by the participant's parent or legal guardian. Adults (participants aged 18 years or older) and older children (participants aged 14-17 years) will self-collect a nasal swab sample by swabbing both nostrils and will test the swab sample themselves on the COVID/Flu Detect™ Rapid Self-Test. For child participants aged 2-13 years, parents or legal guardians will collect a nasal swab sample from their child by swabbing both nostrils and will test the swab sample on behalf of their child on the COVID/Flu Detect™ Rapid Self-Test. The order of collection of the two nasal swab samples will be randomized. A third nasal swab sample may be collected by the participant or the participant's parent, if the first COVID/Flu Detect™ Rapid Self-Test result is invalid. Study staff will observe participants while they self-collect their nasal swab sample and perform the COVID/Flu Detect™ Rapid Self-Test, but participants will not be given any assistance or guidance on these procedures by the study staff.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age, or at least 2 years of age and accompanied by parent or legal guardian.
* Subjects must be willing and able to give informed consent or assent (as age-appropriate).
* Subjects must be able to read/speak English (or Spanish at specific sites) if subject is an adult, minor aged 14 years or older, or parent/guardian of a child subject aged 2 through 13 years.
* Subjects must be currently exhibiting at least two of the following symptoms consistent with possible SARS-CoV-2 or influenza infection: fever or feeling feverish (in absence of documented fever), chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, nasal congestion or runny nose, nausea or vomiting, and/or diarrhea. Subjects must be within 5 days of symptoms onset at enrollment (the day that symptoms start is day 0).

Exclusion Criteria:

* Subject was previously enrolled in this study.
* Subject has undergone a nasal wash or nasal aspirate procedure on day of enrollment.
* Subject has an active nosebleed.
* Subject has received results of an influenza or COVID-19 test within the previous 5 days.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be selected from at least three geographically diverse sites in the United States.
Sampling Method: Probability Sample
Enrollment: 899 (Actual)
Dates: Start 2024-12-26 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
Positive percent agreement (PPA) and negative percent agreement (NPA) of the COVID/Flu Detect™ Rapid Self-Test | Participant samples will be tested on the COVID/Flu Detect™ Rapid Self-Test on the day of enrollment.
  The primary objective of the study is to evaluate the positive percent agreement (PPA) and negative percent agreement (NPA) of the COVID/Flu Detect™ Rapid Self-Test for SARS-CoV-2, influenza A, and influenza B when used in a home-like setting by symptomatic lay users who are within five (5) days of symptoms onset compared to RT-PCR comparator tests for SARS-CoV-2, influenza A, and influenza B. The comparator tests will include an emergency use authorized (EUA) or FDA-cleared SARS-CoV-2 RT-PCR test and an FDA-cleared influenza A and B RT-PCR test.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Cahaba Research, Birmingham, Alabama
  - Medicus Health Research Group Inc, Miami, Florida
  - ASR, LLC, Boise, Idaho
  - Barnes-Jewish Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Ichan School of Medicine at Mount Sinai, Department of Emergency Medicine, New York, New York
  - CHEAR Center LLC., The Bronx, New York
  - Eastside Research Associates, Midland, Texas
  - ERA Health Research, Odessa, Texas

IPD SHARING:
Plan to Share IPD: No